CLINICAL TRIAL: NCT00823602
Title: Comparison Between GnRH Agonist Long Protocol And GnRH Antagonist Protocol In Outcome Of The First Cycle ART
Brief Title: Agonist Gonadotropin-Releasing Hormone (GnRH) Versus Antagonist GnRH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: Razieh Dehghani Firouzabadi, Yazd Research & Clinical Center for Infertility
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1387YAZDRCCI
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Infertility
Keywords: GnRH antagonist; GnRH agonist; pregnancy rate; Ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — ganirelix; Buserelin

ARMS (2):
- 1 (Experimental): GnRH antagonist "ganirelix" 0.25 mg fromm 6th ovarian stimulation
  Interventions: Drug: ganirelix
- 2 (Active Comparator): GnRH agonist, suprefact, stimulation with a standard long protocol
  Interventions: Drug: suprefact

INTERVENTIONS:
Drug: ganirelix — These patients started ovarian stimulation with 150 - 225 IU Gonal F on the second day of menstrual cycle with an S.C. injection once a day. Initiation of 0.25 mg Ganirelix took place on the 6th of the stimulation (fixed protocol) when HMG (Menogon, ferring, pharmacenticals , Germany ).
  Arms: 1
Drug: suprefact — GnRH agonist, standard protocol
  Arms: 2

SUMMARY:
Literature suggests that GnRH antagonists are comparatively more often used in cycles which have an unfavorable prior prognosis, and this protocol is an ideal one for poor responder patients. Up to now, however not enough prospectives have been published to prove any beneficial effect of antagonists on the first cycle assisted reproductive technique.

This prospective study will do to evaluate the efficacy of gonadotropin releasing hormone antagonist in comparison with the standard long protocol in the first cycle of ART.

The investigators will randomize 160 patients undergoing ART for the first time . Group 1 (n=80) was stimulate with a standard long protocol and group 2 (n=80) stimulated with GnRH antagonist and then result of ART compare in two group .

ELIGIBILITY:
Inclusion Criteria:

* first cycle of ART
* age < 35 years
* basal FSH < 10 IU/L

Exclusion Criteria:

* previous IVF or ICSI, hyperprolactinemia, hyperthyroidism, hypothyroidism, uterine abnormality, severe endometriosis
* only one ovary

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 2weeks

SECONDARY OUTCOMES:
ovarian stimulation | 10days

CONTACTS AND LOCATIONS:
Overall Officials: razieh firouzabadi, MD, Study Chair — Yazd Research & Clinical Center for Infertility
Locations (1):
- Yazd Research and Clinical Center For Infertility, Yazd, Yazd Province, Iran